CLINICAL TRIAL: NCT02580097
Title: MR-based Stroke Mechanism and Future Risk Score
Acronym: MR-STARS
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Chief of Radiology, Chinese PLA General Hospital
Other Study IDs: MR-STARS-Radiology-ChinaPLAGH
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Stroke
Keywords: Arterial Spin Labeling; Ischemic stroke; Collateral Circulation; Perfusion imaging
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stroke: Ischemic stroke patients with sympton onset in 24 hours and no contradiction to MRI scan
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI perfusion imaging, including contrast bolus perfusion imaging and arterial spin labeling.

SUMMARY:
To explore prediction model for outcome of patients with acute ischemic stroke using multimodal Magnetic Resonance(MR) imaging was a multicenter prospective observational study supported by National Natural Science Foundation of China. Imaging evaluation of hemodynamic status and antegrade flow were assessed. Patients were followed up to record radiological and clinical outcome. The study recruited patients from 11 centers located in 10 provinces or province-level municipalities across the northeast to the southeast of China mainland.

DETAILED DESCRIPTION:
Patients:

Patients with cerebral ischemia sympton of onset in 24 hours were included. Baseline materials, NIH stroke scale score, modified Rankin Scale at admission, stroke causes, time from sympton onset to enrollment were recorded.

Imaging scan were conducted at admission, within 7 days after admission.

Imaging protocols:

MRI scan protocols: T2 weighted image, T1 weighted image, Diffusion weighted image(DWI), fluid-attenuated inversion recovery(FLAIR), Perfusion weighted image(PWI), arterial spin labeling(ASL) , susceptibility-weighted imaging(SWI).

Contrast agent:

Omniscan 2ml/kg, Inject rate：3ml/s

Digital subtraction angiography(DSA) protocols:

Selective angiography and imaging phase from arterial phase to late venous phase.

Imaging evaluation:

Antegrade flow assessment from ASL Cerebral blood flow(CBF) map. Collateral flow assessment from ASL CBF map, ASL subtraction CBF map, PWI postprocessing map, FLAIR hyperintensity vascular sign.

Initial infarct volume measurement form DWI. Final infarct volume measurement from FLAIR. DWI-ASPECTS. Stroke lesions pattern assessment identified on DWI. DSA antegrade and collateral grade using modified Thrombolysis in Cerebral Infarction(TICI) scale and The American Society of Interventional and Therapeutic Neuroradiology (ASITN) collateral grading system.

Treatment:

Intravenous recombinant tissue plasminogen activator(rtPA), endovascular therapy and conventional treatment including neuro protection, ante-platelet and statin.

Follow up:

within Seven days and a month after imaging follow up and clinical stroke event and modified Rankin Scale(mRS) record in 1 year.

Note:

The original trial from 2015 to 2018 recruited patients with acute and subacute ischemic stroke, and the trial plan was changed to recruit patients with acute cerebral ischemia sympton of onset within 24 h.The study has been upgraded from a single-center study to a multi-center study since 2018.

ELIGIBILITY:
Inclusion Criteria:

* age≥18
* Cerebral ischemic sympton with onset in 24 hours
* pre mRS<2
* All MR examination performed according to study protocol
* Signed informed consent obtained from the patient or patient's legally authorized representative
* Having complete medical history and clinical follow up
* Imaging data can be processed

Exclusion Criteria:

* Intracranial hemorrhage
* Pregnancy and other contraindication to MRI scan
* Informed consent not obtained
* Pre-existing medical, neurological or psychiatric disease that would confound the neurological, functional, or imaging evaluations
* Known allergy to iodine previously refractory to pretreatment medications
* Renal Failure (serum creatinine > 2.0 or Glomerular Filtration Rate [GFR] < 30)
* History of sever kidney disease as an adult, including tumor or transplant surgery, or family history of kidney failure
* Severe cardiac insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients with sympton onset in 24 hours
Sampling Method: Probability Sample
Enrollment: 961 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
modified Rankin Score | Three months
  Modified Rankin Score of patients with acute stroke after 3 months will be followed up for neurological outcome assessment. mRS < 2 is defined as favorable

SECONDARY OUTCOMES:
Final infarct volume | Seven days to 1 month
  Final infarct volume will be measured and infarct volume growth will be calculated.
Stroke event | within 1 year
  The patients will be monitored whether they recured ischemic stroke event including transient ischemic attack (TIA) or stroke confirmed by neurologist and diffusion-weighted image MRI.
mortality | within 1 year
  The patient will be monitored for death by telephone follow-up for neurological outcome assessment

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, M.D.,Ph.D., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lyu J, Xiao S, Meng Z, Wu X, Chen W, Wang G, Niu Q, Li X, Bian Y, Han D, Guo W, Yang S, Bian X, Duan Q, Lan Y, Wang L, Zhang T, Duan C, Chen L, Tian C, Pan Y, Zhou X, Lou X; MR-STARS Investigators. Collateral-Core Ratio as a Novel Predictor of Clinical Outcomes in Acute Ischemic Stroke. Transl Stroke Res. 2023 Feb;14(1):73-82. doi: 10.1007/s12975-022-01066-9. Epub 2022 Jul 25. PMID 35877061